CLINICAL TRIAL: NCT07128238
Title: Research on "Metabolic Adaptation" in Obese People
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SIAT-IRB-250415-H0976
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Body Temperature Changes
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet and Exercise intervention (Experimental): Diet intervention：Provide a fixed amount of food every day Exercise intervention：Train every day according to a specific course schedule
  Interventions: Behavioral: lifestyle intervention

INTERVENTIONS:
Behavioral: lifestyle intervention — This study implemented lifestyle interventions including dietary and exercise interventions. Based on the assessment of the physical condition of the volunteers, a personalized training plan is formulated and a standardized diet is provided. The entire intervention process lasts for 8 weeks.

SUMMARY:
Obesity has become a global public health crisis, with 810 million adults classified as obese (BMI ≥ 30 kg/m²) worldwide in 2020. This number is projected to rise to 1.53 billion by 2035. China faces a particularly severe challenge, with one of the highest rates and fastest growth in obesity prevalence globally. Obesity is a well-established risk factor for numerous chronic diseases, including cancer, cardiovascular disease, and diabetes. As such, weight loss is essential for improving health outcomes and preventing related complications.

Lifestyle interventions-primarily dietary modifications and physical activity-are the cornerstone of obesity treatment, aiming to reduce weight by addressing energy intake and expenditure. Accumulating evidence indicates that energy imbalance is a key driver of obesity. However, resting metabolic rate (RMR), which accounts for approximately 60-75% of total energy expenditure, often declines during lifestyle interventions due to metabolic adaptation. This adaptive decrease in RMR can undermine weight loss efforts.

While both body composition and core body temperature are known to influence RMR, their specific roles in metabolic adaptation during lifestyle interventions remain poorly understood. This study aims to investigate the individual contributions of changes in body composition and fluctuations in core body temperature to the observed reduction in RMR during such interventions. By combining body composition analysis and continuous core temperature monitoring, the study seeks to uncover mechanisms underlying metabolic adaptation and identify potential targets for enhancing weight loss strategies.

DETAILED DESCRIPTION:
Body Composition and Related Measurements Height and Weight Measurement Fasting body weight and height will be measured using the Seca medical metric system (Seca 311231, Germany). Participants will wear a standardized disposable lab coat and stand barefoot on an electronic scale for accurate measurement. Barefoot height will be measured to the nearest millimeter using a Leicester stadiometer (Seca 217, Germany).

3D Body Scanning Participants will stand at the center of the Scanatic™ 360 3D scanning room and maintain proper posture. Trained staff will operate the scanner, sensors, and cameras to collect detailed anthropometric data, including waist and hip circumference.

Bioelectrical Impedance Analysis (BIA) Body composition will be assessed using the TANITA MC-980 device, which provides segmental weight measurements (right arm, left arm, trunk, right leg, left leg) and generates a detailed report including body weight (BW), body fat percentage (fat%), fat mass (FM), body mass index (BMI), and fat-free mass (FFM).

Dual-Energy X-ray Absorptiometry (DXA) DXA scanning (Horizon, Hologic) will be performed with participants wearing uniform disposable lab coats and without metal accessories. DXA uses a low-dose X-ray beam with two energy peaks-one absorbed by soft tissue and the other by bone-to differentiate tissue types. Software algorithms enable precise measurement of fat and fat-free mass.

BOD POD Before testing, participants will fast and avoid strenuous activity, smoking, and exercise for at least two hours. Participants will wear close-fitting swimwear (boxers for men; one-piece swimsuit for women), a swim cap, and no accessories. The BOD POD (GS-X, Cosmed) estimates body composition using air displacement, differentiating fat mass and fat-free mass based on body volume and density calculations.

Magnetic Resonance Imaging (MRI) Whole-body fat distribution will be assessed using the uMR790 MRI system (United Imaging Healthcare). No contrast agent is required. Participants will lie supine on the MRI bed while trained staff perform full-body scans from the neck to the knees using a rapid dynamic imaging sequence. The data will support the development of algorithms for body fat quantification and segmentation.

InBody Analysis InBody provides estimates of body fat percentage, muscle mass, and total body water based on the varying electrical conductivity of different tissues. Participants will stand barefoot and hold electrodes, with hands relaxed. Measurements will be recorded to one decimal place.

Deuterium Dilution Technique Total body water will be measured using the deuterium dilution technique. Participants will fast for 10 hours and provide a baseline urine sample. A dose of deuterium-labeled water (5% deuterium, 95% H₂O) will be administered based on body weight. For example, a 60 kg individual will receive 80.6 g of deuterated water.

Urine samples will be collected at baseline, 3.5 hours post-ingestion, and one week later. Samples will be stored at -20°C and analyzed at the Shenzhen Institutes of Advanced Technology, CAS. Deuterium enrichment typically increases from 150 ppm to 250 ppm and returns to baseline in 14-21 days.

Physical Activity Monitoring (GT3XP-BTLE) Daily activity will be tracked using a tri-axial accelerometer (ActiGraph GT3XP-BTLE, USA), worn continuously except during water-based activities. The device captures physical activity and sleep duration throughout the intervention.

Core Body Temperature Monitoring (e-Celsius) Core temperature will be monitored using the e-Celsius ingestible capsule (BodyCap). The capsule is swallowed under supervision and begins recording temperature approximately 4 hours after ingestion, once it reaches the intestines.

Food Intake Recording Volunteers will record food intake by photographing and weighing their meals. Provided with food scales, they will also use a card-sized object (similar to a bank card) for scale. Photos should include the food before and after eating, along with weight measurements and the card reference.

Metabolic Chamber Total energy expenditure will be measured using a metabolic chamber system (Maastricht Instruments, Netherlands), which operates on indirect calorimetry principles. The system monitors oxygen consumption and CO₂ production continuously over 24 hours. Participants will stay in the chamber from 10 p.m. on Day 1 to 7 a.m. on Day 3.

Breakfast will be provided at 20% of the daily energy requirement, following macronutrient recommendations: protein 15%, fat 25%, and carbohydrates 60%. For lunch and dinner, participants will self-select meals, which will be documented via photographs and weight measurements.

ELIGIBILITY:
Inclusion Criteria:

* BMI： ≥30kg/m2 Willing to participate in an 8-week weight-loss camp program

Exclusion Criteria:

* Metabolic or cardiovascular diseases (such as diabetes) Mental disorders (such as depression and claustrophobia) Infectious diseases (such as AIDS, tuberculosis, malaria) High blood pressure Pregnant, lactating, or prepare for pregnancy Implanted or portable electro-mechanical device Taking antihypertensive or weight-loss medications

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight | About 8 weeks.
  Fasting body weight in kilograms will be measured using the Seca medical metric system (Seca 311231, Germany). Participants will wear a standardized disposable lab coat and stand barefoot on an electronic scale for accurate measurement.
Height | About 8 weeks.
  Height in centimeters will be measured to the nearest millimeter using a Leicester stadiometer (Seca 217, Germany).
Waist circumference | About 8 weeks.
  Waist circumference in centimeters will be measured by 3D Body Scanner. Participants will stand at the center of the ScanatictTM 360 3D scanning room and maintain proper posture. Trained staff will operate the scanner, sensors, and cameras to collect detailed anthropometric data, including waist and hip circumference.
Fat mass | About 8 weeks.
  Fat mass in kilograms will be measured by TANITA MC-980 device and Inbody, which provides segmental weight measurements and generates a detailed report.
Fat-free mass | About 8 weeks.
  Fat-free mass in kilograms will be measured by DXA(Dual-Energy X-ray Absorptiometry). DXA scanning (Horizon, Hologic) will be performed with participants wearing uniform disposable lab coats and without metal accessories.
Fat% | About 8 weeks.
  Fat% will be measured by BOD POD (Air Displacement Plethysmography). Before testing, participants will fast and avoid strenuous activity, smoking, and exercise for at least two hours. Participants will wear close-fitting swimwear (boxers for men; one-piece swimsuit for women), a swim cap, and no accessories. The BOD POD (GS-X, Cosmed) estimates body composition using air displacement, differentiating fat mass and fat-free mass based on body volume and density calculations.
Total body volume | About 8 weeks.
  Total body volume in liters will be measured by MRI (United Imaging uMR790). Whole-body fat distribution will be assessed using the uMR790 MRI system (United Imaging Healthcare). No contrast agent is required. Participants will lie supine on the MRI bed while trained staff perform full-body scans from the neck to the knees using a rapid dynamic imaging sequence.
Total body water | About 7 days.
  Total body water in kilograms will be measured by deuterium dilution technique. Participants will fast for 10 hours and provide a baseline urine sample. A dose of deuterium-labeled water (5%deuterium, 95% H2O) will be administered based on body weight. For example, a 60 kg individual will receive 80.6 g of deuterated water.
  Urine samples will be collected at baseline, 3.5 hours post-ingestion, and one week later. Samples will be stored at -20℃ and analyzed at the Shenzhen Institutes of Advanced Technology, CAS. Deuterium enrichment typically increases from 150 ppm to 250 ppm and returns to baseline in 14-21 days.
Physical Activity | About 10 weeks.
  Daily activity will be tracked using a tri-axial accelerometer (ActiGraph GT3XP- BTLE, USA), worn continuously except during water-based activities. The device captures physical activity and sleep duration throughout the intervention.
Core Body Temperature | About 3 days.
  Core body temperature in degree centigrade will be measured by the e-Celsius ingestible capsule (BodyCap). The capsule is swallowed uner supervision and begins recording temperature approximately 4 hours after ingestion, once it reaches the intestines.
Food Intake | About 8 weeks.
  Food intake in grams will be measured by food scales. Volunteers will record food intake by photographing and weighing their meals. Provided with food scales, they will also use a card-sized object (similar to a bank card) for scale. Photos should include the food before and after eating, along with weight measurements and the card reference.
Total energy expenditure | About 3 days.
  Total energy expenditure will be measured using a metabolic chamber system (Maastricht Instruments, Netherlands), which operates on indirect calorimetry principles. The system monitors oxygen consumption and CO2 production continuously over 24 hours. Participants will stay in the chamber from 10 p.m. on Day 1 to 7 a.m. on Day 3.
  Breakfast will be provided at 20% of the daily energy requirement, following macronutrient recommendations: protein 15%, fat 25%, and carbohydrates 60%. For lunch and dinner, participants will self-select meals, which will be documented via photographs and weight measurements.